CLINICAL TRIAL: NCT00534313
Title: A Phase IIB, Multi-Dose, Multi-center, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Abatacept Versus Placebo in the Treatment of Psoriatic Arthritis
Brief Title: Safety and Efficacy of Abatacept Versus Placebo in Participants With Psoriatic Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy with respect to skin-related lesions in the short-term phase
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM101-158; EUDRACT 2007-004241-15
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Results first posted 2010-11-22 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Abatacept (30/10) (Active Comparator): Abatacept (30 mg/kg) was administered as intravenous (iv) infusion over approximately 30 minutes on Days 1 and 15, followed by 10 mg/kg (fixed dose) abatacept infusion on Day 29 and every 28 days thereafter up to and including Day 141. The dose was calculated based on screening visit weight of participants for dosing on Days 1 and 15 followed by fixed dosing as per rheumatoid arthritis label (participants weighing <60 kg received 500 mg, participants weighing 60 to 100 kg received 750 mg, and participants weighing >100 kg received 1000 mg) thereafter.
  Interventions: Drug: Abatacept
- Abatacept (10/10) (Active Comparator): Abatacept (10 mg/kg) was administered as iv infusion over approximately 30 minutes on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141 in the double-blind period and continued for next 18 months in the open-label period till Day 729. All participants received a dose based on their screening visit weight as per rheumatoid arthritis label (participants weighing <60 kg received 500 mg, participants weighing 60 to 100 kg received 750 mg, and participants weighing >100 kg received 1000 mg).
  Interventions: Drug: Abatacept
- Abatacept (3/3) (Active Comparator): Abatacept (3 mg/kg) was administered as iv infusion over approximately 30 minutes on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141. The dose was calculated based on screening visit weight of participants.
  Interventions: Drug: Abatacept
- Placebo (Placebo Comparator): Placebo solution (5% dextrose in water for injection, 0.9% sodium chloride injection) by iv infusion was administered on Days 1, 15, and 29 and every 28 days thereafter till Day 141.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Abatacept — Solution, intravenous, monthly, short-term = 24 weeks (6 months)
  Other Names: Orencia; BMS-188667
  Arms: Abatacept (10/10); Abatacept (3/3); Abatacept (30/10)
Drug: Placebo — Solution, intravenous, placebo (double dummy), monthly, short-term = 24 weeks (6 months)
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine an optimal abatacept dosing regimen for the treatment of active arthritis due to psoriatic arthritis in patients who have had a prior inadequate response to disease-modifying antirheumatic drugs, including methotrexate and tumor necrosis factor alpha-blockade compounds.

ELIGIBILITY:
Key Inclusion Criteria:

* Meeting classification criteria for psoriatic arthritis for a duration of disease of at least 3 months
* Prior failure (inefficacy or intolerance) of therapy with disease-modifying antirheumatic drugs; if patient had prior failure of methotrexate, he or she must have been taking at least 15 mg per week for at least 2 months
* If recent failure(inefficacy or intolerance) of a tumor necrosis factor α-blockade compound, participant must be washed out prior to first dose: 56 days for infliximab and 28 days for etanercept and adalimumab
* Disease activity as defined by a tender joint count of ≥3, swollen joint count of ≥3, and clinically detectable synovitis at screening and Day 01 (prior to infusion)
* Active psoriasis with a qualifying target lesion ≥2 cm in diameter
* Able to undergo magnetic resonance imaging
* Use of appropriate birth control by women of child bearing potential (WOCBP)

Key Exclusion Criteria:

* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 10 weeks after the last dose of investigational product
* Women who are pregnant or breastfeeding or who plan to become pregnant or to start breastfeeding during the duration of the study
* Women with a positive pregnancy test on enrollment or prior to investigational product administration.
* Participants scheduled for or anticipating joint replacement surgery.
* Those with a recent history of clinically significant drug or alcohol abuse
* Concomitant illness that in the investigator's opinion is likely to require systemic glucocorticosteroid therapy during the study (for example: moderate to severe asthma)
* Current symptoms of severe, progressive, or uncontrolled renal, hepatic, hematologic, pulmonary, cardiac, neurologic, ophthalmologic, or cerebral disease.
* Unwillingness or inability to undergo screening based on current local or country guidelines/standards to evaluate the presence of cancer
* Cancer within the last 5 years
* Current malignancy or signs of possible malignancy detected by screening procedures for which the workup to exclude malignancy has not been completed or malignancy cannot be excluded
* At risk for or history (within 3 years) of tuberculosis
* Any serious bacterial infection within the last 3 months, not treated and resolved with antibiotics, or any chronic bacterial infection (such as, but not limited to, chronic pyelonephritis, osteomyelitis, and bronchiectasis)
* Evidence of active or latent bacterial or viral infection infections at the time of potential enrollment
* Herpes zoster or cytomegalovirus resolving less than 2 months prior to signing informed consent
* Receipt of any live vaccines within 3 months of the anticipated first dose of study medication or anticipation of the need for a live vaccine at any time during and for 3 months after the duration of the study

Long-term period participants: Must have met eligibility criteria for short-term period and completed short-term (24-week) period of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (44):
- United States (19):
  - Rheumatology Associates Of North Alabama, Huntsville, Alabama
  - Desert Medical Advances, Palm Desert, California
  - Stanford University School Of Medicine, Palo Alto, California
  - Boling Clinical Trials, Upland, California
  - Joao Nascimento, Bridgeport, Connecticut
  - New England Research Associates, Llc, Trumbull, Connecticut
  - Sarasota Arthritis Research Center, Sarasota, Florida
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Justus Fiechtner, Md, Mph, Lansing, Michigan
  - St. Paul Rheumatology P.A., Eagan, Minnesota
  - Midwest Arthritis Center, Kalamazoo, Minnesota
  - Arthritis Clinic & Carolina Bone & Joint, Pa, Charlotte, North Carolina
  - Deaconess Hospital, Cincinnati, Ohio
  - Health Research Of Oklahoma, Oklahoma City, Oklahoma
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Rheumatic Disease Associates, Ltd., Willow Grove, Pennsylvania
  - Chase, Walter F., Austin, Texas
  - Seattle Rheumatology Associates, Seattle, Washington
  - Arthritis Northwest, Spokane, Washington
- Argentina (3):
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, Santa Fe, Santa Fe Province
- Australia (3):
  - Local Institution, Cairns, Queensland
  - Local Institution, Maroochydore, Queensland
  - Local Institution, Fitzroy, Melbourne, Victoria
- Belgium (2):
  - Local Institution, Hasselt
  - Local Institution, Leuven
- Canada (4):
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, Montreal, Quebec
  - Local Institution, Québec, Quebec
  - Local Institution, Trois-Rivières, Quebec
- France (3):
  - Local Institution, Chambray-lès-Tours
  - Local Institution, Lille
  - Local Institution, Montpellier
- Germany (3):
  - Local Institution, Frankfurt am Main
  - Local Institution, Hamburg
  - Local Institution, Hildesheim
- Italy (3):
  - Local Institution, Napoli
  - Local Institution, Potenza
  - Local Institution, Reggio Emilia
- Local Institution, Amsterdam, Netherlands
- Local Institution, Lillehammer, Norway
- Local Institution, Panorama, Western Cape, South Africa
- Local Institution, A Coruña, Spain

REFERENCES:
- [Derived] Ostergaard M, Bird P, Pachai C, Du S, Wu C, Landis J, Fuerst T, Ahmad HA, Connolly SE, Conaghan PG. Implementation of the OMERACT Psoriatic Arthritis Magnetic Resonance Imaging Scoring System in a randomized phase IIb study of abatacept in psoriatic arthritis. Rheumatology (Oxford). 2022 Nov 2;61(11):4305-4313. doi: 10.1093/rheumatology/keac073. PMID 35137002
- [Derived] Mease P, Genovese MC, Gladstein G, Kivitz AJ, Ritchlin C, Tak PP, Wollenhaupt J, Bahary O, Becker JC, Kelly S, Sigal L, Teng J, Gladman D. Abatacept in the treatment of patients with psoriatic arthritis: results of a six-month, multicenter, randomized, double-blind, placebo-controlled, phase II trial. Arthritis Rheum. 2011 Apr;63(4):939-48. doi: 10.1002/art.30176. PMID 21128258

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 191 participants were enrolled and 21 were not randomized. Reasons for this included: adverse events (AEs) (2); participant withdrew consent (5); lost to follow up (1); participant no longer meets study criteria (13).
Groups:
- Abatacept 30/10: Participants were administered intravenous (iv) infusions of abatacept (30 mg/kg - calculated dose) over approximately 30 minutes on Days 1 and 15, followed by 10 mg/kg (fixed dose) abatacept infusion on Day 29 and every 28 days thereafter up to and including Day 141. All participants received a calculated dose on Day 1 and 15 followed by fixed dose based on their screening visit weight i.e. for participants weighing < 60 kg received 500 mg, participants weighing 60 kg to 100 kg received 750 mg and participants weighing > 100 kg received 1000 mg.
- Abatacept 10/10: Participants were administered iv infusions of abatacept (10 mg/kg) over approximately 30 minutes on Days 1, 15, 29 and every 28 days thereafter up to and including Day 141. All participants received a dose based on their screening visit weight as per rheumatoid arthritis label (participants weighing < 60 kg received 500 mg, participants weighing 60 kg to 100 kg received 750 mg and participants weighing > 100 kg received 1000mg).
- Abatacept 3/3: Participants were administered iv infusions of abatacept (3 mg/kg - calculated dose) over approximately 30 minutes on Days 1, 15, 29 and every 28 days thereafter up to and including Day 141. All participants received calculated dose based on their screening visit weight.
- Placebo: Participants were administered iv infusions of either dextrose 5% solution or 0.9% sodium chloride solution at a constant rate over approximately 30 minutes on Days 1, 15, 29 and every 28 days thereafter up to and including Day 141.
Period: Short-term Period
Arm/Group | Abatacept 30/10 | Abatacept 10/10 | Abatacept 3/3 | Placebo
Started | 43 | 40 | 45 | 42
Completed | 37 (Completed the short-term study) | 34 (Completed the short-term study) | 43 (Completed the short-term study) | 33 (Completed the short-term study)
Not Completed | 6 | 6 | 2 | 9
Not completed — Adverse Event | 1 | 2 | 1 | 3
Not completed — Lack of Efficacy | 3 | 4 | 0 | 3
Not completed — Participant not meeting study criteria | 0 | 0 | 0 | 1
Not completed — Participant withdrew consent | 2 | 0 | 0 | 2
Not completed — Pregnancy | 0 | 0 | 1 | 0
Period: Long-term Period
Arm/Group | Abatacept 30/10 | Abatacept 10/10 | Abatacept 3/3 | Placebo
Started | 37 | 34 | 43 | 33
Completed | 0 | 0 | 0 | 0
Not Completed | 37 | 34 | 43 | 33
Not completed — Adverse Event | 2 | 1 | 0 | 1
Not completed — Lack of Efficacy | 14 | 10 | 14 | 12
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 0
Not completed — No longer meets study criteria | 0 | 1 | 0 | 0
Not completed — Poor compliance/noncompliance | 0 | 1 | 1 | 0
Not completed — Administrative reason by sponsor | 17 | 15 | 26 | 18
Not completed — Other | 1 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abatacept 30/10 | Abatacept 10/10 | Abatacept 3/3 | Placebo | Total
Number analyzed (Participants) | 43 | 40 | 45 | 42 | 170
Age Continuous [Median (Full Range); unit: years] | 54.0 [29.0 to 69.0] | 51.5 [26.0 to 73.0] | 51.0 [29.0 to 72.0] | 53.0 [30.0 to 82.0] | 52.0 [26.0 to 82.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 14 | 23 | 19 | 79
  Male | 20 | 26 | 22 | 23 | 91
Race/Ethnicity, Customized [Number; unit: participants]
  White | 43 | 38 | 44 | 41 | 166
  Asian | 0 | 2 | 1 | 0 | 3
  Pacific | 0 | 0 | 0 | 1 | 1
Weight [Mean (Standard Deviation); unit: kilograms] | 92.9 (21.3) | 85.0 (17.9) | 85.0 (19.1) | 96.0 (19.4) | 89.7 (19.9)

OUTCOME MEASURES:

1. Primary Outcome: Long-term Period: Number of Participants With Death As Outcome, Serious Adverse Events (SAEs), Drug-related SAEs, SAEs Leading to Discontinuation, Adverse Events (AEs), Drug-related AEs, AEs Leading to Discontinuation, and AEs of Interest
Description: Presp=prespecified; acute= ≤1 hour after start of infusion; periinfusional= ≤24 hours after start of infusion. AE=any new unfavorable symptom or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=an unfavorable medical event that at any dose results in death, significant disability, drug dependency/abuse, hospitalization or prolonged hospitalization; is life-threatening, an important medical event, or a congenital anomaly/birth defect. Drug-related=possibly, probably, or certainly related and of unknown relationship to study drug.
Time Frame: From Day 169 to Day 729
Population: All participants who received at least 1 infusion of abatacept during the long-term period.
Measure: Number; unit: Participants
Groups:
- All Treated Participants: Long-term period: All participants received an open-label abatacept weight-tiered dose of 10 mg/kg at Day 169 and every 28 days.
Arm/Group | All Treated Participants
Number analyzed (Participants) | 147
Participants
  Deaths | 0
  SAEs | 20
  Drug-related SAEs | 4
  SAEs leading to discontinuation | 0
  AEs | 123
  Drug-related AEs | 58
  AES leading to discontinuation | 4
  AEs of Interest (AEI): Infections | 83
  AEI: Malignancy | 2
  AEI: Autoimmune disorders (presp) | 5
  AEI: Infusion reactions (presp): Acute | 4
  AEI: Infusion reactions (presp): Periinfusional | 11

2. Secondary Outcome: Long-term Period: Percentage of Participants Achieving American College of Rheumatology (ACR) 20, ACR 50, ACR 70, ACR 90 Responses at Days 365 and 729
Description: An ACR 20 (50, 70, 90) responder was a participant whose counts for both tender and swollen joints was reduced by 20% (50%, 70%, 90%, respectively) or more from baseline and who had a reduction of 20% (50%, 70%, 90%, respectively) or more from baseline in 3 of the following assessments: participant's assessment of disease activity, participant's global assessment of disease activity, Investigators Global Response, participant's assessment of physical function by Health Assessment Questionnaire Disability Index, and Disease Activity Score 28 based on C-reactive protein.
Time Frame: At Days 365 and 729 from Baseline
Population: All participants who received at least 1 infusion of abatacept in the long-term (open-label) period. (n=number of participants with a response)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Abatacept 30/10: Short-term period: Participants received IV infusions of abatacept (30 mg/kg, calculated-dose) over approximately 30 minutes on Days 1 and 15, followed by 10 mg/kg (fixed-dose) abatacept infusion on Day 29 and every 28 days thereafter up to and including Day 141. All participants received a calculated dose on Days 1 and 15 followed by fixed dose based on their screening visit weight (participants weighing <60 kg received 500 mg, 60 to 100 kg received 750 mg, and >100 kg received 1000 mg. Long-term period: Participants received an open-label abatacept weight-tiered dose of 10 mg/kg at Day 169 and every 28 days.
- Abatacept 10/10: Short-term period: Participants received IV infusions of abatacept (10 mg/kg) over approximately 30 minutes on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141. All participants received a dose based on their screening visit weight as per rheumatoid arthritis label (participants weighing <60 kg received 500 mg, 60 to 100 kg received 750 mg, and >100 kg received 1000 mg). Long-term period: Participants received an open-label abatacept weight-tiered dose of 10 mg/kg at Day 169 and every 28 days.
- Abatacept 3/3: Short-term period: Participants received IV infusions of abatacept (3 mg/kg, calculated-dose) over approximately 30 minutes on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141. All participants received calculated dose based on their screening visit weight. Long-term period: Participants received an open-label abatacept weight-tiered dose of 10 mg/kg at Day 169 and every 28 days.
- Placebo: Short-term period: Participants received IV infusions of either dextrose 5% solution or 0.9% sodium chloride solution at a constant rate over approximately 30 minutes on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141. Long-term period: Participants received an open-label abatacept weight-tiered dose of 10 mg/kg at Day 169 and every 28 days.
Arm/Group | Abatacept 30/10 | Abatacept 10/10 | Abatacept 3/3 | Placebo
Number analyzed (Participants) | 37 | 34 | 43 | 33
Percentage of participants
  ACR 20, Day 365 (n=34, 29, 36, 32) | 50.0 [33.2 to 66.8] | 62.1 [44.4 to 79.7] | 61.1 [45.2 to 77.0] | 46.9 [29.6 to 64.2]
  ACR 20, Day 729 (n=21, 18, 26, 18) | 81 [64.2 to 97.7] | 66.7 [44.9 to 88.4] | 65.4 [47.1 to 83.7] | 72.2 [51.5 to 92.9]
  ACR 50, Day 365 (n=34, 29, 36, 32) | 23.5 [9.3 to 37.8] | 37.9 [20.3 to 55.6] | 33.3 [17.9 to 48.7] | 34.4 [17.9 to 50.8]
  ACR 50, Day 729 (n=21, 18, 26, 18) | 57.1 [36.0 to 78.3] | 27.8 [7.1 to 48.5] | 42.3 [23.3 to 61.3] | 55.6 [32.6 to 78.5]
  ACR 70, Day 365 (n=34, 29, 36, 32) | 5.9 [0.0 to 13.8] | 17.2 [3.5 to 31.01] | 13.9 [2.6 to 25.2] | 18.8 [5.2 to 32.2]
  ACR 70, Day 729 (n=21, 18, 26, 18) | 23.8 [5.6 to 42.0] | 16.7 [0.0 to 33.9] | 23.1 [6.9 to 39.3] | 11.1 [0.0 to 25.6]
  ACR 90, Day 365 (n=34, 29, 36, 32) | 0 [0.0 to 0.0] | 6.9 [0.0 to 16.1] | 5.6 [0.0 to 13.0] | 6.3 [0.0 to 14.6]
  ACR 90, Day 729 (n=21, 18, 26, 18) | 0 [0.0 to 0.0] | 5.6 [0.0 to 16.1] | 11.5 [0.0 to 23.8] | 0 [0.0 to 0.0]

3. Secondary Outcome: Long-term Period: Number of Participants With an Investigators Global Assessment (IGA) Score of Clear or Almost Clear at Days 365 and 729
Description: IGA score indicates lesion induration, scaling, and erythema: 0=clear (no signs of plaque psoriasis except for residual discoloration); 1=almost clear (just perceptible erythema, no induration to very slightly elevated above normal skin levels, limited amount of very fine scaling); 2=mild disease (mild erythema, mild induration, mainly fine scaling predominates); 3=moderate disease (moderate erythema [most plaques are red], moderate induration and/or coarse scale predominates); 4=severe (severe erythema, marked to very marked elevation of lesions, coarse thick scale predominates).
Time Frame: From Day 169 to Days 365 and 729
Population: as for outcome 2
Measure: Number; unit: Participants
Groups:
- Abatacept 10/10: Short-term period: Participants received IV infusions of abatacept (10 mg/kg) over approximately 30 minutes on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141. All participants received a dose based on their screening visit weight as per rheumatoid arthritis label (participants weighing <60 kg received 500 mg, 60 to 100 kg received 750 mg, and >100 kg received 1000 mg).Long-term period: participants received an open-label abatacept weight-tiered dose of 10 mg/kg at Day 169 and every 28 days.
- Abatacept 3/3: Short-term period: Participants received IV infusions of abatacept (3 mg/kg, calculated-dose) over approximately 30 minutes on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141. All participants received calculated dose based on their screening visit weight.Long-term period: participants received an open-label abatacept weight-tiered dose of 10 mg/kg at Day 169 and every 28 days.
Arm/Group | Abatacept 30/10 | Abatacept 10/10 | Abatacept 3/3 | Placebo
Number analyzed (Participants) | 37 | 34 | 43 | 33
Participants
  Day 365 (n=30, 29, 34, 23) | 13 | 10 | 19 | 10
  Day 729 (n=20, 17, 26, 18) | 10 | 7 | 16 | 8

4. Secondary Outcome: Long-term Period: Mean Percentage of Change From Baseline in Target Lesion Score at Days 365 and 729
Description: Target lesion score is a measurement of the degree of erythema, induration, and scale of a psoriatic lesion, at least 2 cm in diameter, selected as a target for response throughout the study period. The scores assigned were 0=clear, 1=almost clear, 2=mild clear, 3=moderate disease, 4=severe. Percent improvement from baseline was computed using the ratio of improvement from baseline to the baseline value.
Time Frame: From Baseline to Days 365 and 729
Population: All participants who received at least 1 infusion of abatacept in the long-term (open-label) period.
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Abatacept 30/10 | Abatacept 10/10 | Abatacept 3/3 | Placebo
Number analyzed (Participants) | 37 | 34 | 43 | 33
Percentage of change
  Day 365 | 27.51 (7.92) | 41.97 (7.90) | 20.32 (8.59) | 33.82 (7.52)
  Day 729 | 49.14 (9.13) | 45.07 (7.98) | 44.79 (9.09) | 34.41 (8.98)

5. Secondary Outcome: Long-term Period: Mean Change From Baseline in the Short-form 36 (SF-36), Version 2, Domain and Component Scores at Days 365 and 729
Description: PCS=physical component score; MCS=mental component score. The SF-36 is a 36-item instrument with physical and mental components and covers quality of life (QoL) domains: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. Responses are used to derive physical and mental component summary scores, ranging from 0 to 100, with higher scores indicating better QoL. Mean change from baseline=postbaseline value-baseline value; a higher value signifies improvement.
Time Frame: At Days 365 and 729 from baseline
Measure: Mean (Standard Error); unit: Units on a scale
Groups:
- Abatacept 30/10: Short-term period: Participants received intravenous (IV) infusions of abatacept (30 mg/kg, calculated-dose) over approximately 30 minutes on Days 1 and 15, followed by 10 mg/kg (fixed-dose) abatacept infusion on Day 29 and every 28 days thereafter up to and including Day 141. All participants received a calculated dose on Days 1 and 15 followed by fixed dose based on their screening visit weight (participants weighing <60 kg received 500 mg, 60 to 100 kg received 750 mg, and >100 kg received 1000 mg. Long-term period: participants received an open-label abatacept weight-tiered dose of 10 mg/kg at Day 169 and every 28 days.
Arm/Group | Abatacept 30/10 | Abatacept 10/10 | Abatacept 3/3 | Placebo
Number analyzed (Participants) | 37 | 34 | 43 | 33
Units on a scale
  Day 365 PCS (n=34, 32, 37,29) | 1.73 (1.10) | 7.59 (1.36) | 4.86 (1.67) | 3.59 (1.19)
  Day 365 MCS (n=34,32, 37,29) | 2.73 (1.60) | 1.07 (2.00) | 4.95 (2.10) | 4.40 (2.00)
  Day 729 PCS (n=20,18, 26,18) | 5.59 (1.43) | 7.97 (2.0) | 6.74 (1.95) | 4.45 (1.14)
  Day 729 MCS (n=20,18, 26,18) | 5.89 (1.84) | -0.17 (2.71) | 1.85 (2.11) | 4.35 (2.29)

6. Secondary Outcome: Long-term Period: Number of Participants Achieving A Reduction of At Least 0.3 Unit From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Days 365 and 729
Description: Per the HAQ-DI, participants assessed their own ability to perform the following tasks: dress/groom, arise, eat, walk, reach, grip, maintain hygiene, and maintain daily activity over a period by marking their responses on a questionnaire. Scoring of the HAQ-DI: 0=without any difficulty; 1=with some difficulty; 2=with much difficulty); and 3=unable to do. Greater score=greater disability. Responders with a >= 0.3 unit decrease in index scores from baseline to days 365 and 729 were considered to be improved.
Time Frame: Days 365 and 729 from baseline
Population: All participants who received at least 1 infusion of abatacept in the long-term (open-label) period. (n=number of participants with responses available)
Measure: Number; unit: Participants
Arm/Group | Abatacept 30/10 | Abatacept 10/10 | Abatacept 3/3 | Placebo
Number analyzed (Participants) | 37 | 34 | 43 | 33
Participants
  Day 365 (n=3, 28, 32, 23) | 12 | 16 | 17 | 12
  Day 729 (n=9, 11, 13, 10) | 9 | 11 | 13 | 10

7. Secondary Outcome: Short-term Period: Number of Participants With Marked Abnormalities in Hematology
Description: LLN=lower limit of normal; ULN=upper limit of normal; pre-Rx=pretreatment. Marked abnormalities are laboratory measurements marked as abnormal, per predefined study criteria, at any study time point. Criteria: Hemoglobin >3 g/dL decrease from pre-Rx value; hematocrit <0.75*pre-Rx value; erythrocytes <0.75*pre-Rx value; platelets <0.67*LLN (or, if pre-Rx value <LLN, <0.5*pre-Rx value and <100000/mm^3) or >1.5*ULN.
Time Frame: From Baseline to Day 169
Population: All participants who received at least 1 infusion of study medication during double-blind period. n=number of participants with evaluable results (each arm respectively).
Measure: Number; unit: Participants
Groups:
- Abatacept 30/10: Participants received iv infusions of abatacept (30 mg/kg - calculated dose) over approximately 30 minutes on Days 1 and 15, followed by 10 mg/kg (fixed dose) abatacept infusion on Day 29 and every 28 days thereafter up to and including Day 141. All participants received a calculated dose on Day 1 and 15 followed by fixed dose based on their screening visit weight (participants weighing <60 kg received 500 mg, participants weighing 60 to 100 kg received 750 mg, and participants weighing >100 kg received 1000 mg.
- Abatacept 10/10: Participants received iv infusions of abatacept (10 mg/kg) over approximately 30 minutes on Days 1, 15,and 29 and every 28 days thereafter up to and including Day 141. All participants received a dose based on their screening visit weight as per rheumatoid arthritis label (participants weighing <60 kg received 500 mg, participants weighing 60 to 100 kg received 750 mg and participants weighing >100 kg received 1000 mg).
- Placebo: Participants received iv infusions of either dextrose 5% solution or 0.9% sodium chloride solution at a constant rate over approximately 30 minutes on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141.
Arm/Group | Abatacept 30/10 | Abatacept 10/10 | Abatacept 3/3 | Placebo
Number analyzed (Participants) | 43 | 40 | 45 | 42
Participants
  Hemoglobin (n = 43, 40, 45, 41) | 0 | 0 | 0 | 0
  Hematocrit (n = 43, 40, 45, 41) | 0 | 0 | 0 | 0
  Erythrocytes (n = 43, 40, 45, 41) | 0 | 0 | 0 | 0
  Platelet count (n = 43, 40, 45, 41) | 0 | 0 | 0 | 0

8. Primary Outcome: Short-term Period: Number of Participants With ACR 20 Response at Day 169
Description: An ACR 20 responder was a participant who had a reduction of 20% or more from baseline in scores for both tender and swollen joints and had a reduction from baseline of 20% or more in 3 out of the following 5 assessments: participant's assessment of disease activity, participant's global assessment of disease activity, investigator's global assessment of disease activity, participant's assessment of physical function by HAQ-DI, and Disease Activity Score 28-C reactive protein.
Time Frame: At Day 169 from Baseline
Population: All randomized participants who received at least 1 infusion of study medication in the double-blind (short-term) period. Missing response values were imputed as nonresponders for participants who discontinued early after receiving study medication.
Measure: Number; unit: Participants
Groups:
- Abatacept 30/10: Short-term period: Participants received intravenous (IV) infusions of abatacept (30 mg/kg, calculated-dose) over approximately 30 minutes on Days 1 and 15, followed by 10 mg/kg (fixed-dose) abatacept infusion on Day 29 and every 28 days thereafter up to and including Day 141. All participants received a calculated dose on Days 1 and 15 followed by fixed dose based on their screening visit weight (participants weighing <60 kg received 500 mg, 60 to 100 kg received 750 mg, and >100 kg received 1000 mg.
- Abatacept 10/10: Short-term period: Participants received IV infusions of abatacept (10 mg/kg) over approximately 30 minutes on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141. All participants received a dose based on their screening visit weight as per rheumatoid arthritis label (participants weighing <60 kg received 500 mg, 60 to 100 kg received 750 mg, and >100 kg received 1000 mg).
- Abatacept 3/3: Short-term period: Participants received IV infusions of abatacept (3 mg/kg, calculated-dose) over approximately 30 minutes on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141. All participants received calculated dose based on their screening visit weight.
- Placebo: Short-term period: Participants received IV infusions of either dextrose 5% solution or 0.9% sodium chloride solution at a constant rate over approximately 30 minutes on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141.
Arm/Group | Abatacept 30/10 | Abatacept 10/10 | Abatacept 3/3 | Placebo
Number analyzed (Participants) | 43 | 40 | 45 | 42
Participants | 18 | 19 | 15 | 8
Statistical Analysis 1: Comparison: Abatacept 30/10 vs Placebo; Test type: Superiority or Other; p = 0.022, Cochran-Mantel-Haenszel — The p-value (two-sided) was based on Cochran-Mantel-Haenszel method (CMH) with stratification of baseline body surface area (BSA) affected by psoriasis; Difference = 22.9, 95% CI 2-sided [4.0 to 41.8] — Difference was based on CMH with stratification of baseline BSA affected by psoriasis
Statistical Analysis 2: Comparison: Abatacept 10/10 vs Placebo; Test type: Superiority or Other; p = 0.006, Cochran-Mantel-Haenszel — p-value (two-sided) was based on CMH with stratification of baseline BSA affected by psoriasis; Difference = 28.7, 95% CI 2-sided [9.4 to 48.0] — Difference was based on CMH with stratification of baseline BSA affected by psoriasis
Statistical Analysis 3: Comparison: Abatacept 3/3 vs Placebo; Test type: Superiority or Other; p = 0.121, Cochran-Mantel-Haenszel — p-value (2-sided) was based on CMH with stratification of baseline BSA affected by psoriasis; Difference = 14.6, 95% CI 2-sided [-3.5 to 32.6] — Difference was based on CMH with stratification of baseline BSA affected by psoriasis

9. Secondary Outcome: Short-term Period: Number of Participants With Marked Abnormalities in Hematology (Continued)
Description: LLN=lower limit of normal; ULN=upper limit of normal; pre-Rx=pretreatment. Laboratory measurements are marked as abnormal per predefined study criteria, at any study time point. Criteria for the data presented. Leukocytes <0.75*LLN or >1.25*ULN (or, if pre-Rx value <LLN, <0.8*pre-Rx or >ULN. If pre-Rx value >ULN, >1.2*pre-Rx or <LLN); neutrophils+bands (absolute) <1.00*10^3 c/uL; lymphocytes (absolute) <0.75*10^3 c/uL or >7.50*10^3 c/uL; monocytes (absolute) >2000/mm^3; basophils (absolute) >0.40*10^3 c/uL; eosinophils (absolute) >0.75*10^3 c/uL.
Time Frame: From Baseline to Day 169
Population: as for outcome 7
Measure: Number; unit: Participants
Groups:
- Abatacept 30/10: Participants who received iv infusions of abatacept (30 mg/kg-calculated dose) over approximately 30 minutes on Days 1 and 15, followed by 10 mg/kg (fixed dose) abatacept infusion on Day 29 and every 28 days thereafter up to and including Day 141. All participants received a calculated dose on Day 1 and 15 followed by fixed dose based on their screening visit weight (participants weighing <60 kg received 500 mg, participants weighing 60 to 100 kg received 750 mg, and participants weighing >100 kg received 1000 mg.
- Abatacept 10/10: Participants received iv infusions of abatacept (10 mg/kg) over approximately 30 minutes on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141. All participants received a dose based on their screening visit weight as per rheumatoid arthritis label (participants weighing <60 kg received 500 mg, participants weighing 60 kg to 100 kg received 750 mg, and participants weighing >100 kg received 1000 mg).
- Abatacept 3/3: Participants received iv infusions of abatacept (3 mg/kg - calculated dose) over approximately 30 minutes on Days 1, 15, 29 and every 28 days thereafter up to and including Day 141. All participants received calculated dose based on their screening visit weight.
Arm/Group | Abatacept 30/10 | Abatacept 10/10 | Abatacept 3/3 | Placebo
Number analyzed (Participants) | 43 | 40 | 45 | 42
Participants
  Leukocytes (n = 43, 40, 45, 41) | 0 | 0 | 2 | 0
  Neutrophils+bands (absolute) (n = 43, 40, 45, 41) | 0 | 0 | 0 | 0
  Lymphocytes (absolute) (n = 43, 40, 45, 41) | 2 | 0 | 6 | 1
  Monocytes (absolute) (n = 43, 40, 45, 41) | 0 | 0 | 0 | 0
  Basophils (absolute) (n = 43, 40, 45, 41) | 0 | 0 | 0 | 0
  Eosinophils (absolute) (n = 43, 40, 45, 41) | 1 | 1 | 1 | 0

10. Secondary Outcome: Short-term Period: Number of Participants With Marked Abnormalities in Serum Chemistry
Description: ULN=upper limit of normal; pre-Rx=pretreatment. Marked abnormality criteria: Alkaline phosphatase (ALP), gamma-glutamyltransferase (GGT) >2*ULN (if pre-Rx >ULN, >3*pre-Rx); aspartate aminotransferase (AST), alanine transaminase (ALT) >3*ULN (if pre-Rx >ULN, >4*pre-Rx); bilirubin (total) >2*ULN (if pre-Rx >ULN, >4*pre-Rx); blood urea nitrogen (BUN) >2*pre-Rx; creatinine >1.5*pre-Rx.
Time Frame: Baseline to Day 169
Population: All participants who received at least 1 infusion of study medication during the double-blind period. n=number of participants with evaluable results (each arm respectively).
Measure: Number; unit: Participants
Groups:
- Abatacept 30/10: Participants received iv infusions of abatacept (30 mg/kg - calculated dose) over approximately 30 minutes on Days 1 and 15, followed by 10 mg/kg (fixed dose) abatacept infusion on Day 29 and every 28 days thereafter up to and including Day 141. All participants received a calculated dose on Days 1 and 15 followed by fixed dose based on their screening visit weight (participants weighing <60 kg received 500 mg, participants weighing 60 to 100 kg received 750 mg, and participants weighing >100 kg received 1000 mg.
- Abatacept 10/10: Participants received iv infusions of abatacept (10 mg/kg) over approximately 30 minutes on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141. All participants received a dose based on their screening visit weight as per rheumatoid arthritis label (participants weighing <60 kg received 500 mg, participants weighing 60 to 100 kg received 750 mg, and participants weighing >100 kg received 1000 mg).
- Abatacept 3/3: Participants received iv infusions of abatacept (3 mg/kg - calculated dose) over approximately 30 minutes on Days 1, 15,and 29 and every 28 days thereafter up to and including Day 141. All participants received calculated dose based on their screening visit weight.
Arm/Group | Abatacept 30/10 | Abatacept 10/10 | Abatacept 3/3 | Placebo
Number analyzed (Participants) | 43 | 40 | 45 | 42
Participants
  ALP (n = 43, 40, 45, 41) | 0 | 0 | 0 | 0
  AST (n = 43, 40, 45, 41) | 0 | 0 | 0 | 0
  ALT (n = 43, 40, 45, 41) | 1 | 0 | 0 | 0
  GGT (n = 43, 40, 45, 41) | 1 | 0 | 0 | 0
  Bilirubin (total) (n = 43, 40, 45, 41) | 0 | 0 | 0 | 0
  BUN (n = 43, 40, 45, 41) | 0 | 0 | 0 | 0
  Creatinine (n = 43, 40, 45, 41) | 0 | 0 | 0 | 0

11. Secondary Outcome: Short-term Period: Number of Participants With Marked Abnormalities in Serum Chemistry (Continued)
Description: LLN=lower limit of normal; ULN=upper limit of normal; pre-Rx=pretreatment. Marked abnormality criteria: Sodium <0.95*LLN or >1.05*ULN (if pre-Rx<LLN, <0.95*pre-Rx or >ULN. If pre-Rx >ULN,>1.05* pre-Rx or <LLN); potassium, chloride <0.9*LLN or >1.1*ULN (if pre-Rx <LLN, <0.9*pre-Rx or >ULN. If pre-Rx >ULN, >1.1*pre-Rx or <LLN); calcium <0.8*LLN or >1.2*ULN (if pre-Rx <LLN,<0.75* pre-Rx or >ULN. If pre-Rx >ULN, >1.25* pre-Rx or <LLN); phosphorous <0.75*LLN or >1.25*ULN (if pre-Rx <LLN, <0.67*pre-Rx or >ULN. If pre-Rx >ULN, >1.33*pre-Rx or <LLN.
Time Frame: Baseline to Day 169
Population: as for outcome 10
Measure: Number; unit: Participants
Groups:
- Abatacept 10/10: Participants received iv infusions of abatacept (10 mg/kg) over approximately 30 minutes on Days 1, 15,and 29 and every 28 days thereafter up to and including Day 141. All participants received a dose based on their screening visit weight as per rheumatoid arthritis label (participants weighing <60 kg received 500 mg, participants weighing 60 to 100 kg received 750 mg, and participants weighing >100 kg received 1000 mg).
- Abatacept 3/3: Participants received iv infusions of abatacept (3 mg/kg - calculated dose) over approximately 30 minutes on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141. All participants received calculated dose based on their screening visit weight.
Arm/Group | Abatacept 30/10 | Abatacept 10/10 | Abatacept 3/3 | Placebo
Number analyzed (Participants) | 43 | 40 | 45 | 42
Participants
  Sodium (n = 43, 40, 45, 41) | 0 | 0 | 0 | 0
  Potassium (n = 43, 40, 45, 41) | 0 | 0 | 0 | 1
  Chloride (n = 43, 40, 45, 41) | 0 | 0 | 0 | 0
  Calcium (total) (n = 43, 40, 45, 41) | 0 | 0 | 0 | 0
  Phosphorous , inorganic (n = 43, 40, 45, 41) | 0 | 0 | 1 | 1

12. Secondary Outcome: Short-term Period: Number of Participants With Marked Abnormalities in Serum Chemistry (Continued)
Description: LLN=lower limit of normal; ULN=upper limit of normal; pre-Rx=pretreatment. Marked abnormality criteria: Glucose <65 or >220 mg/dL; glucose (fasting)<0.8*LLN or >1.5*ULN (if pre-Rx <LLN, <0.8*pre-Rx or >ULN. If pre-Rx >ULN, t>2.0*pre-Rx or <LLN). Protein (total) <0.9*LLN or >1.1*ULN (if pre-Rx <LLN, <0.9*pre-Rx or >ULN. If pre-Rx >ULN, >1.1*pre-Rx or <LLN). Albumin <0.9*LLN (if pre-Rx <LLN, <0.75* pre-Rx). Uric acid >1.5*ULN; if pre-Rx >ULN or >2*pre-Rx value.
Time Frame: From Baseline to Day 169
Population: All participants who received at least 1 infusion of study medication during the double-blind period. n=number of participants with evaluable results.
Measure: Number; unit: Participants
Arm/Group | Abatacept 30/10 | Abatacept 10/10 | Abatacept 3/3 | Placebo
Number analyzed (Participants) | 43 | 40 | 45 | 42
Participants
  Glucose (n = 43, 40, 45, 41) | 1 | 4 | 8 | 2
  Glucose, fasting (n = 16, 12, 12, 15) | 0 | 0 | 0 | 0
  Protein (total) (n = 43, 40, 45, 41) | 0 | 0 | 0 | 0
  Albumin (n = 43, 40, 45, 41) | 0 | 0 | 0 | 0
  Uric acid (n = 43, 40, 45, 41) | 0 | 0 | 0 | 0

13. Secondary Outcome: Short-term Period: Number of Participants With Marked Abnormalities in Urinalysis
Description: Pre-Rx=pretreatment. Criteria for marked abnormality: Protein, glucose, blood, leukocyte esterase, red blood cells (RBC), white blood cells (WBC) >=2+ (or, if value >=4, or if pre-Rx value=0 or 0.5, >= 2* or if pre-RX value =1, >=3, or if pre-Rx =2 or 3, >=4).
Time Frame: From Baseline to Day 169
Population: All participants who received at least 1 infusion of study medication during the double-blind period. n = number of participants with evaluable results (each arm respectively).
Measure: Number; unit: Participants
Groups:
- Placebo: Participants received iv infusions of either dextrose 5% solution or 0.9% sodium chloride solution at a constant rate over approximately 30 minutes on Days 1, 15,and 29 and every 28 days thereafter up to and including Day 141.
Arm/Group | Abatacept 30/10 | Abatacept 10/10 | Abatacept 3/3 | Placebo
Number analyzed (Participants) | 43 | 40 | 45 | 42
Participants
  Protein (n = 42, 37, 38, 40) | 0 | 0 | 0 | 1
  Glucose (n = 42, 37, 38, 40) | 0 | 0 | 0 | 1
  Blood (n = 42, 37, 38, 40) | 2 | 2 | 3 | 2
  Leukocyte esterase (n = 3, 7, 4, 5) | 0 | 0 | 1 | 1
  WBC (n = 6, 8, 8, 6) | 1 | 1 | 3 | 3
  RBC (n = 6, 7, 5, 6) | 3 | 1 | 1 | 2

14. Secondary Outcome: Short-term Period: Number of Participants Who Died and With SAEs, AEs, AEs Leading to Discontinuation, SAEs Leading to Discontinuation, Drug-related AEs, and Drug-related SAEs
Description: An AE is any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not necessarily have a causal relationship with treatment. An SAE is any unfavorable medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency or abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Drug-related=possibly, probably, or certainly related to and of unknown relationship to study treatment.
Time Frame: From Baseline to Day 169
Population: All participants who received at least 1 infusion of study medication during the double-blind period.
Measure: Number; unit: Participants
Arm/Group | Abatacept 30/10 | Abatacept 10/10 | Abatacept 3/3 | Placebo
Number analyzed (Participants) | 43 | 40 | 45 | 42
Participants
  Deaths | 0 | 0 | 0 | 0
  SAEs | 4 | 2 | 0 | 1
  AEs | 29 | 31 | 31 | 30
  All AEs Leading to Discontinuation | 1 | 2 | 1 | 3
  All SAEs Leading to Discontinuation | 1 | 0 | 0 | 0
  Drug-related AEs | 13 | 13 | 12 | 7
  Drug-related SAEs | 1 | 1 | 0 | 0

15. Secondary Outcome: Short-term Period: Number of Participants With an IGA Score of Clear or Almost Clear at Day 169
Description: Score indicates lesion induration, scaling, and erythema: 0 = clear (no signs of plaque psoriasis except for residual discoloration); 1 = almost clear (just perceptible erythema, no induration to very slightly elevated above normal skin levels, limited amount of very fine scaling); 2 = mild disease (mild erythema, mild induration, mainly fine scaling predominates); 3 = moderate disease (moderate erythema [most plaques are red], moderate induration and/or coarse scale predominates); 4=severe (severe erythema, marked to very marked elevation of lesions, coarse thick scale predominates).
Time Frame: At Day 169 from Baseline
Population: All randomized participants who received at least 1 infusion of study medication in double-blind (short-term) period. Missing response values were imputed as nonresponders for participants who discontinued early after receiving study medication.
Measure: Number; unit: Participants
Groups:
- Abatacept 30/10: Short-term period: Participants received IV infusions of abatacept (30 mg/kg, calculated-dose) over approximately 30 minutes on Days 1 and 15, followed by 10 mg/kg (fixed-dose) abatacept infusion on Day 29 and every 28 days thereafter up to and including Day 141. All participants received a calculated dose on Days 1 and 15 followed by fixed dose based on their screening visit weight (participants weighing <60 kg received 500 mg, 60 to 100 kg received 750 mg, and >100 kg received 1000 mg.
Arm/Group | Abatacept 30/10 | Abatacept 10/10 | Abatacept 3/3 | Placebo
Number analyzed (Participants) | 43 | 40 | 45 | 42
Participants | 9 | 10 | 17 | 11
Statistical Analysis 1: Comparison: Abatacept 30/10 vs Placebo; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Difference = -6.0, 95% CI 2-sided [-23.0 to 11.0] — Difference and 95% confidence intervals (CI) was based on CMH with stratification of baseline BSA affected by psoriasis
Statistical Analysis 2: Comparison: Abatacept 10/10 vs Placebo; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Difference = -0.5, 95% CI 2-sided [-18.0 to 17.1] — Difference and 95% CI was based on CMH with stratification of baseline BSA affected by psoriasis
Statistical Analysis 3: Comparison: Abatacept 3/3 vs Placebo; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Difference = 10.4, 95% CI 2-sided [-7.6 to 28.5] — Difference and 95% CI was based on CMH with stratification of baseline BSA affected by psoriasis

16. Secondary Outcome: Short-term Period: Mean Percentage of Change From Baseline in Target Lesion Score at Day 169
Description: Target lesion score measures the degree of erythema, induration, and scale of a psoriatic lesion with a diameter of at least 2 cm, selected as a target for response throughout the study period. Scores: 0=clear, 1=almost clear, 2=mild clear, 3=moderate disease, 4=severe. Percent improvement from baseline was computed using the ratio of improvement from baseline to the baseline value.
Time Frame: At Day 169 from Baseline
Population: All randomized participants who received at least 1 infusion of study drug in double-blind (short-term) period. Only participants with both baseline and postbaseline values included. Missing values at Day 169 were imputed using the last observation carried forward values, except for participants with only baseline value.
Measure: Mean (Standard Error); unit: Percentage of change
Groups:
- Abatacept 30/10: Participants received iv infusions of abatacept (30 mg/kg - calculated dose) over approximately 30 minutes on Days 1 and 15, followed by 10 mg/kg (fixed dose) abatacept infusion on Day 29 and every 28 days thereafter up to and including Day 141. All participants received a calculated dose on Days 1 and 15 followed by fixed dose based on their screening visit weight (participants weighing <60 kg received 500 mg, participants weighing 60 to 100 kg received 750 mg, and participants weighing >100 kg received 1000 mg).
- Abatacept 3/3: Participants received iv infusions of abatacept (3 mg/kg - calculated dose) over approximately 30 minutes on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141. All participants received a calculated dose based on their screening visit weight.
Arm/Group | Abatacept 30/10 | Abatacept 10/10 | Abatacept 3/3 | Placebo
Number analyzed (Participants) | 43 | 40 | 45 | 42
Percentage of change | 19.39 (9.16) | 22.96 (9.46) | 31.11 (8.98) | 0.63 (9.35)
Statistical Analysis 1: Comparison: Abatacept 30/10 vs Placebo; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 18.77, 95% CI 2-sided [-7.02 to 44.56]
Statistical Analysis 2: Comparison: Abatacept 10/10 vs Placebo; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 22.34, 95% CI 2-sided [-3.93 to 48.60]
Statistical Analysis 3: Comparison: Abatacept 3/3 vs Placebo; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 30.48, 95% CI 2-sided [4.82 to 56.15]

17. Secondary Outcome: Short-term Period: Number of Participants With Positive Responses for Serum Levels of Abatacept-specific Antibodies (Anti-Abatacept-C)
Description: Meso Scale Discovery electrochemiluminescence, a validated, sensitive immunoassay technique (anti-abatacept assay C) was used to measure serum levels of abatacept-specific antibodies against the whole molecule (both the CTLA4 and possibly immunoglobulin G portion [anti-abatacept antibody].
Time Frame: From Baseline to Day 169
Population: Participants who received abatacept and for whom baseline and at least 1 additional measurement were available during the double-blind (short-term) period.
Measure: Number; unit: Participants
Groups:
- Abatacept 10/10: Participants received iv infusions of abatacept (10 mg/kg) over approximately 30 minutes on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 169. All participants received a dose based on their screening visit weight as per by rheumatoid arthritis label (participants weighing <60 kg received 500 mg, participants weighing 60 to 100 kg received 750 mg, and participants weighing >100 kg received 1000mg).
Arm/Group | Abatacept 30/10 | Abatacept 10/10 | Abatacept 3/3
Number analyzed (Participants) | 43 | 40 | 45
Participants | 1 | 0 | 2

18. Secondary Outcome: Short-term Period: Mean Change From Baseline in the Mental Component Summary Score as Measured by the Short-form 36 at Day 169
Description: PCS=physical component score; MCS=mental component score. The Short-form 36 is a 36-item instrument with physical and mental components and covers quality of life (QoL) domains: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. Responses are used to derive physical and mental component summary scores, ranging from 0 to 100, with higher scores indicating better QoL. Mean change from baseline=postbaseline value-baseline value; a higher value signifies improvement.
Time Frame: At Day 169 from Baseline
Population: All randomized and treated participants with baseline and postbaseline measurements at Day 169. Missing values were imputed by Last Observation Carried Forward, except for participants with only baseline observations.
Measure: Mean (Standard Error); unit: Units on a scale
Groups:
- Abatacept 30/10: Participants received calculated dose) over approximately 30 minutes on Days 1 and 15, followed by 10 mg/kg (fixed dose) abatacept infusion on Day 29 and every 28 days thereafter up to and including Day 141. All participants received a calculated dose on Days 1 and 15 followed by fixed dose based on their screening visit weight (participants weighing <60 kg received 500 mg, participants weighing 60 to 100 kg received 750 mg and participants weighing >100 kg received 1000 mg.
- Abatacept 10/10: Participants received iv infusions of abatacept (10 mg/kg) over approximately 30 minutes on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141. All participants received a dose based on their screening visit weight as per rheumatoid arthritis label (participants weighing < 60 kg received 500 mg, participants weighing 60 kg to 100 kg received 750 mg and participants weighing > 100 kg received 1000mg).
Arm/Group | Abatacept 30/10 | Abatacept 10/10 | Abatacept 3/3 | Placebo
Number analyzed (Participants) | 42 | 40 | 43 | 41
Units on a scale | 4.50 (2.45) | 4.42 (2.50) | 3.16 (2.41) | 2.41 (2.47)
Statistical Analysis 1: Comparison: Abatacept 30/10 vs Placebo; Test type: Superiority or Other; ANCOVA; ANCOVA model with treatment as factor and baseline value as covariate was used for the analysis; Mean Difference (Net) = 2.08, 95% CI [-4.79 to 8.96]
Statistical Analysis 2: Comparison: Abatacept 10/10 vs Placebo; Test type: Superiority or Other; ANCOVA; ANCOVA model with treatment as factor and baseline value as covariate was used for the analysis; Mean Difference (Net) = 2.01, 95% CI 2-sided [-4.94 to 8.95]
Statistical Analysis 3: Comparison: Abatacept 3/3 vs Placebo; Test type: Superiority or Other; ANCOVA; ANCOVA model with treatment as factor and baseline value as covariate was used for the analysis; Mean Difference (Net) = 0.75, 95% CI 2-sided [-6.08 to 7.58]

19. Secondary Outcome: Short-term Period: Mean Serum Concentrations of Abatacept
Description: Abatacept was assayed using a validated enzyme linked immunosorbent assay method (ELISA). Serum concentration versus time data was analyzed in the descriptive pharmacokinetic (PK) analysis.
Time Frame: Days 1, 15, 29, 57, 85, 113, 141, and 169
Population: All participants who received at least 1 infusion of study medication and were evaluable for PK analysis during double-blind period. n= number of participants with evaluable PK results in each arm respectively.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Abatacept 30/10 | Abatacept 10/10 | Abatacept 3/3
Number analyzed (Participants) | 43 | 40 | 45
µg/mL
  Day 1 (n= 13, 13, 44) | 0 (0) | 0.01 (0.01) | 0 (0)
  Day 15 (n= 43, 38, 42) | 119.99 (35.30) | 48.29 (17.96) | 14.28 (7.67)
  Day 29 (n= 41, 39, 43) | 186.82 (62.49) | 49.70 (16.79) | 16.20 (4.86)
  Day 57 (n= 40, 39, 44) | 58.55 (26.09) | 25.75 (9.67) | 10.42 (5.75)
  Day 85 (n= 37, 35, 41) | 39.00 (19.37) | 26.29 (10.59) | 8.73 (3.26)
  Day 113 ( n= 35, 33, 43) | 36.30 (19.94) | 32.69 (14.08) | 8.85 (5.01)
  Day 141 (n= 35, 34, 42) | 26.70 (9.24) | 25.78 (9.74) | 7.66 (3.13)
  Day 169 (n= 36, 42, 34) | 28.93 (11.29) | 26.34 (10.75) | 9.29 (5.23)

20. Secondary Outcome: Short-term Period: Mean Serum Trough Concentrations (Cmin) of Abatacept
Description: Abatacept was assayed using a validated ELISA method. Cmin of abatacept was obtained from concentration versus time data.
Time Frame: Days 1, 15, 29, 57, 85, 113, 141, and 169
Population: as for outcome 19
Measure: Geometric Mean (Full Range); unit: µg/mL
Groups:
- Abatacept 10/10: Participants received iv infusions of abatacept (10 mg/kg) over approximately 30 minutes on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141. All participants received a dose based on their screening visit weight as per rheumatoid arthritis label (participants weighing <60 kg received 500 mg, participants weighing 60 to 100 kg received 750 mg, and participants weighing >100 kg received 1000mg).
Arm/Group | Abatacept 30/10 | Abatacept 10/10 | Abatacept 3/3
Number analyzed (Participants) | 43 | 40 | 45
µg/mL
  Day 15 (n= 43, 38, 43) | 115.35 [70.65 to 236.39] | 45.10 [21.27 to 95.96] | 12.81 [4.25 to 39.81]
  Day 29 (n= 41, 39, 43) | 176.22 [68.45 to 373.07] | 46.86 [21.23 to 87.55] | 15.43 [4.99 to 28.15]
  Day 57 (n= 40, 39, 44) | 53.08 [11.21 to 151.10] | 23.88 [8.18 to 50.84] | 9.03 [2.53 to 33.88]
  Day 85 (n= 37, 35, 41) | 33.09 [1.87 to 94.46] | 24.36 [10.47 to 55.13] | 8.15 [2.97 to 16.01]
  Day 113 (n= 35, 33, 43) | 31.50 [8.30 to 78.91] | 29.60 [6.66 to 71.21] | 7.56 [2.14 to 27.82]
  Day 141 (n= 35, 34, 42) | 25.02 [10.77 to 43.31] | 23.62 [7.24 to 45.66] | 6.91 [1.50 to 14.32]
  Day 169 (n= 36, 34, 42) | 26.65 [10.05 to 53.77] | 24.33 [11.65 to 50.31] | 7.84 [1.68 to 28.85]

21. Secondary Outcome: Short-term Period: Population Pharmacokinetic (POPPK) Analysis of the Pharmacokinetic (PK) Parameters
Description: PK data: summaries of concentrations and concentration versus time plots were obtained. These data were to be used to develop a POPPK model using a nonlinear mixed-effects model. Prediction of PK data for each of the 3 abatacept treatment groups using POPPK methodology was not performed, because it would not provide any relevant information over the observed PK data.
Time Frame: Days 1, 15, 29, 57, 85, 113, 141, and 169
Arm/Group | Abatacept 30/10 | Abatacept 10/10 | Abatacept 3/3 | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

22. Secondary Outcome: Short-term Period: Mean Change From Baseline in Physical Component Summary Score as Measured by the Short-form 36 at Day 169
Description: as for outcome 18
Time Frame: At Day 169 from Baseline
Population: All randomized participants who received treatment and with baseline and postbaseline measurements at Day 169. Missing values were imputed by Last Observation Carried Forward, except for participants with only baseline observations.
Measure: Mean (Standard Error); unit: Units on a scale
Groups:
- Abatacept 30/10: Participants received iv infusions of abatacept (30 mg/kg -calculated dose) over approximately 30 minutes on Days 1 and 15, followed by 10 mg/kg (fixed dose) abatacept infusion on Day 29 and every 28 days thereafter up to and including Day 141. All participants received a calculated dose on Days 1 and 15 followed by fixed dose based on their screening visit weight (participants weighing <60 kg received 500 mg, participants weighing 60 to 100 kg received 750 mg, and participants weighing >100 kg received 1000 mg.
Arm/Group | Abatacept 30/10 | Abatacept 10/10 | Abatacept 3/3 | Placebo
Number analyzed (Participants) | 42 | 40 | 43 | 41
Units on a scale | 7.30 (1.85) | 9.27 (1.91) | 6.32 (1.82) | 0.15 (1.87)
Statistical Analysis 1: Comparison: Abatacept 30/10 vs Placebo; Test type: Superiority or Other; ANCOVA; Analysis of covariance (ANCOVA) model with treatment as factor and baseline value as covariate was used for the analysis; Mean Difference (Net) = 7.15, 95% CI 2-sided [1.97 to 12.33]
Statistical Analysis 2: Comparison: Abatacept 10/10 vs Placebo; Test type: Superiority or Other; ANCOVA; ANCOVA model with treatment as factor and baseline value as covariate was used for the analysis; Mean Difference (Net) = 9.12, 95% CI 2-sided [3.83 to 14.41]
Statistical Analysis 3: Comparison: Abatacept 3/3 vs Placebo; Test type: Superiority or Other; ANCOVA; ANCOVA model with treatment as factor and baseline value as covariate was used for the analysis; Mean Difference (Net) = 6.17, 95% CI 2-sided [1.01 to 11.32]

23. Secondary Outcome: Short-term Period: Number of Participants Achieving a Reduction of At Least 0.3 Unit From Baseline in HAQ-DI Scores at Day 169
Description: The HAQ-DI assesses a participant's ability to perform the following tasks: dress/groom; arise; eat; walk; reach; grip; maintain hygiene; and maintain daily activity over a period by marking their response on a questionnaire. Responses/scores range from: 0=without any difficulty, 1=with some difficulty, 2=with much difficulty, 3=to unable to do. Higher total score=greater disability.
Time Frame: At Day 169 from Baseline
Population: All randomized participants who received at least 1 infusion of study medication at any time. Missing response values were imputed as nonresponders for participants who discontinued early after receiving study medication.
Measure: Number; unit: Participants
Groups:
- Abatacept 10/10: Participants received iv infusions of abatacept (10 mg/kg) over approximately 30 minutes on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141. All participants received a dose based on their screening visit weight as per rheumatoid arthritis label (participants weighing <60 kg received 500 mg, participants weighing 60 to 100 kg received 750 mg and participants weighing >100 kg received 1000mg).
Arm/Group | Abatacept 30/10 | Abatacept 10/10 | Abatacept 3/3 | Placebo
Number analyzed (Participants) | 43 | 40 | 45 | 42
Participants | 15 | 18 | 16 | 8
Statistical Analysis 1: Comparison: Abatacept 30/10 vs Placebo; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Difference = 16.0, 95% CI 2-sided [-2.5 to 34.5] — Difference and 95% CI was based on CMH with stratification of baseline BSA affected by psoriasis
Statistical Analysis 2: Comparison: Abatacept 10/10 vs Placebo; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Difference = 26.1, 95% CI [6.8 to 45.5] — Difference and 95% CI was based on CMH with stratification of baseline BSA affected by psoriasis
Statistical Analysis 3: Comparison: Abatacept 3/3 vs Placebo; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Difference = 16.6, 95% CI [-1.8 to 34.9] — Difference and 95% CI was based on CMH with stratification of baseline BSA affected by psoriasis

ADVERSE EVENTS:
Groups:
- Abatacept 10/10 (Short-term Period): Participants received IV infusions of abatacept (10 mg/kg) over approximately 30 minutes on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141. All participants received a dose based on their screening visit weight as per rheumatoid arthritis label (participants weighing <60 kg received 500 mg, 60 to 100 kg received 750 mg, and >100 kg received 1000 mg).
- Abatacept 3/3 (Short-term Period): Participants received IV infusions of abatacept (3 mg/kg, calculated-dose) over approximately 30 minutes on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141. All participants received calculated dose based on their screening visit weight.
- Abatacept 30/10 (Short-term Period): Participants received IV infusions of abatacept (30 mg/kg, calculated-dose) over approximately 30 minutes on Days 1 and 15, followed by 10 mg/kg (fixed-dose) abatacept infusion on Day 29 and every 28 days thereafter up to and including Day 141. All participants received a calculated dose on Days 1 and 15 followed by fixed dose based on their screening visit weight (participants weighing <60 kg received 500 mg, 60 to 100 kg received 750 mg, and >100 kg received 1000 mg.
- Abatacept (Long-term Period): Participants received an open-label abatacept weight-tiered dose of 10 mg/kg at Day 169 and every 28 days.
- Placebo (Short-term Period): Participants received IV infusions of either dextrose 5% solution or 0.9% sodium chloride solution at a constant rate over approximately 30 minutes on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141.
Arm/Group | Abatacept 10/10 (Short-term Period) | Abatacept 3/3 (Short-term Period) | Abatacept 30/10 (Short-term Period) | Abatacept (Long-term Period) | Placebo (Short-term Period)
Serious Adverse Events (participants affected / at risk) | 2/40 | 1/45 | 4/43 | 20/147 | 1/42
Other Adverse Events (participants affected / at risk) | 16/40 | 15/45 | 16/43 | 73/147 | 19/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept 10/10 (Short-term Period) (N=40) | Abatacept 3/3 (Short-term Period) (N=45) | Abatacept 30/10 (Short-term Period) (N=43) | Abatacept (Long-term Period) (N=147) | Placebo (Short-term Period) (N=42)
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 2 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Lentigo maligna stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Personality disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Family stress (Social circumstances) | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept 10/10 (Short-term Period) (N=40) | Abatacept 3/3 (Short-term Period) (N=45) | Abatacept 30/10 (Short-term Period) (N=43) | Abatacept (Long-term Period) (N=147) | Placebo (Short-term Period) (N=42)
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0 | 8 | 2
Nausea (Gastrointestinal disorders) | 2 | 1 | 2 | 6 | 3
Chest pain (General disorders) | 1 | 0 | 1 | 10 | 1
Fatigue (General disorders) | 3 | 1 | 1 | 3 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 3 | 13 | 1
Nasopharyngitis (Infections and infestations) | 4 | 5 | 4 | 33 | 4
Sinusitis (Infections and infestations) | 2 | 1 | 2 | 12 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 2 | 16 | 2
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 10 | 0
Headache (Nervous system disorders) | 1 | 3 | 4 | 9 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 8 | 1
Hypertension (Vascular disorders) | 3 | 1 | 1 | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.